CLINICAL TRIAL: NCT02861846
Title: Predictive Value of Biomarkers of the Alzheimer's Disease (AD) in Elderly Patients With New-onset Epilepsy
Acronym: BIOMALEPSIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL16-0041; 2016-A00563-48 (Other: ID-RCB)
Record Dates: First submitted 2016-07-04; First posted 2016-08-10 (Estimated); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Epilepsy
Keywords: epilepsy; Alzheimer; biomarkers; predictive value
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Presence of biomarkers of AD in cerebrospinal fluid (Other): Patients older than 60 years, with normal brain MRI and with normal cognitive functioning who demonstrate a profile of CSF biomarkers of AD suggestive of biological AD
  Interventions: Biological: profile of CSF biomarkers of AD

INTERVENTIONS:
Biological: profile of CSF biomarkers of AD — dosage of biomarker of AD

SUMMARY:
Beyond 60 years, the prevalence of epilepsy is estimated at approximately 1% and increases with age. In these patients, the etiology of epilepsy is unknown in 25% of cases, even up to 55% after 65 years. Although new-onset epilepsy in the elderly is associated with a vascular disease in 50% of cases, the hypothesis of an ongoing neurodegenerative process, including an Alzheimer's disease (AD), is also common. However, investigators do not have any marker that might help to identify the patients who develop epilepsy after 60 years and who might be, despite a normal cognitive functioning, already engaged in the pathophysiological process of AD.

A number of data suggest a link between the pathophysiological process of AD and epileptogenesis:

(i) a third of patients with epilepsy develops MA, (ii) the occurrence of epilepsy in AD is an aggravating factor for cognition, (iii) in animal models of AD, the relationship between neuronal hyperexcitability and amyloid deposits is bidirectional, the amyloid protein has a pro-seizure effect and the presence of epilepsy increases the amyloid deposits, (iv) in these models, the administration of an antiepileptic drug protects from deterioration of cognition, (v) the close relationship between amyloid and neuronal hyperexcitability might be mediated by the inflammatory processes associated with AD, and particularly the microglial activation which role in epileptogenesis has been shown elsewhere.

Investigators hypothesize that in a subgroup of patients who develop epilepsy after 60 years, the occurrence of epilepsy might reflect the presence of an ongoing amyloid pathology. Our goal is to identify through biomarkers of AD in the cerebrospinal fluid of patients who develop an epilepsy after 60 years with normal MRI and normal cognition those at high risk of later developing clinically defined AD.

Identifying patients with amyloid pathology which would be expressed through epilepsy before the onset of cognitive dysfunction might help to adapt both the management of seizures and of the cognitive dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years
* Patients with newly diagnosed epilepsy according to the latest criteria of the International League against Epilepsy.
* MMSE ≥ 28/30.
* Patients with or without cognitive complaints.
* Patients whose brain MRI did not reveal significant abnormalities outside slight cortical atrophy.
* Patients in whom the lumbar puncture did not revealed abnormalities suggestive of an infectious disease or a limbic encephalitis.
* Patient with adequate visual and auditory skills, an oral and written language in French available to clinical and neuropsychological assessment.
* Patient who have given its written consent.

Exclusion Criteria:

* Previous history of epilepsy before age 60 years.
* Patient with against-indication to MRI (pacemaker, ferromagnetic clips, mechanical heart valves, intra-cochlear implants, intraocular foreign body, skin or other) or refusing MRI.
* Presence of an abnormality in brain MRI.
* Patients with diagnostic criteria for dementia of Alzheimer's disease, vascular dementia, mixed dementia or frontotemporal lobar degeneration.
* Patients with autoimmune encephalitis.
* Patients under legal protection measure

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2023-03-16 (Actual); Study Completion 2023-03-16 (Actual)

PRIMARY OUTCOMES:
The primary endpoint was the number of patients in a population of subjects older than 60 years with new-onset epilepsy but without cognitive impairment whose profile of the CSF biomarkers of the AD is suggestive of an AD. | 2 years

SECONDARY OUTCOMES:
changes in episodic verbal memory at 2 years | 2 years
  Evolution of RL/RI-16 score between inclusion and 2 years of follow-up
changes in visual recognition memory at 2 years | 2 years
  Evolution of DMS 48 score between inclusion and 2 years of follow-up
Evolution of DO 80 score | 2 years
  Evolution of semantic memory at 2 years: Evolution of DO 80 score between inclusion and 2 years follow-up
Evolution of categorical influences | 2 years
  Evolution of semantic memory at 2 years: Evolution of categorical influences between inclusion and 2 years follow-up
Evolution of TOP 10 score | 2 years
  Evolution of semantic memory at 2 years: Evolution of TOP 10 score between inclusion and 2 years follow-up
Changes in monthly frequency of seizures at 2 years | 2 years
  Evolution of monthly frequency of seizures between inclusion and 2 years of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Aurélie RICHARD-MORNAS, Doctor, Study Director — Hospices Civils de Lyon
Locations (4):
- France (4):
  - Hospices Civils de Lyon, Bron
  - CHU Gabriel- Montpied, Clermont-Ferrand
  - CHU des Alpes, Grenoble
  - CHU Hôpital Nord, Saint-Etienne

IPD SHARING:
Plan to Share IPD: Undecided